CLINICAL TRIAL: NCT02474394
Title: The Comparison of the Effects of McGrath Video Laryngoscope and the Macintosh Laryngoscope on Intraocular Pressure: A Randomized Trial
Brief Title: Effects of Videolaryngoscope on Intraocular Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, M.D., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IOP-1
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Intubation Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mcgrath (Active Comparator): The endotracheal intubation will be provided using Mcgrath series 5 video laryngoscope
  Interventions: Device: Mcgrath
- Macintosh (Active Comparator): The endotracheal incubation will be provided using macintosh laryngoscope
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Mcgrath — The patient will be intubated using McGrath series 5 video laryngoscope and the intraocular pressure of the patient will be evaluated with Tonopen XL tonometer
  Other Names: videolaryngoscope
  Arms: Mcgrath
Device: Macintosh — The patient will be intubated using Macintosh laryngoscope and the intraocular pressure of the patient will be evaluated with Tonopen XL tonometer
  Other Names: Conventional Laryngoscope
  Arms: Macintosh

SUMMARY:
This study is designed to compare the effects of the McGrath Series 5 video laryngoscope and Macintosh laryngoscope on intraocular pressure during laryngoscopy.

DETAILED DESCRIPTION:
The stability of the intraocular pressure plays an important role during ophthalmic surgery. The systemic blood pressure, aqueous humor dynamics, choroidal blood volume, central venous pressure, extra-ocular muscle tone, and also conventional laryngoscopy affect the intraocular pressure.It was shown that the new devices for laryngoscopy, such as video laryngoscopes provide minimal hemodynamic changes when compared to direct laryngoscopes. However there is no current data about the effects of the intubation with McGrath videolaryngoscope on intraocular pressure. The main objective of this study to compare the effects of the McGrath Series 5 video laryngoscope and Macintosh laryngoscope on intraocular pressure during laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist physical status I
* Non-ophthalmic elective surgery under general anesthesia

Exclusion Criteria:

* A history of pre-existing glaucoma or previous intraocular surgery
* Thyromental distance below 6cm
* Maximum mouth opening below 3cm
* Mallampati score of III or IV
* Pre-anesthetic intraocular pressure above 20 mmHg
* Number of intubation attempts more than 2
* Obstetric or laparoscopic surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | during laryngoscopy
  The intraocular pressure measurement will be performed using a Tono-Pen XL tonometer (Reichert Inc., USA) by an ophthalmologist who is blind to the intubation device used.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaman, M.D., Principal Investigator — Gaziosmanpasa University Medical School
Locations (1):
- Gaziosmanpasa University Medical School, Tokat Province, Turkey (Türkiye)